CLINICAL TRIAL: NCT04821622
Title: TALAPRO-3: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, STUDY OF TALAZOPARIB WITH ENZALUTAMIDE VERSUS PLACEBO WITH ENZALUTAMIDE IN MEN WITH DDR GENE MUTATED METASTATIC CASTRATION-SENSITIVE PROSTATE CANCER
Brief Title: Study of Talazoparib With Enzalutamide in Men With DDR Gene Mutated mCSPC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3441052; TALAPRO-3 (Other: Alias Study Number); 2024-510809-28-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: DDR; prostate cancer; castration-sensitive; PARP-inhibitor; hormone-sensitive; metastatic hormone-sensitive prostate cancer; Advanced prostate cancer; Metastatic castration-sensitive prostate cancer; mCSPC; enzalutamide; metastatic prostate cancer; DNA Damage Response; DNA Damage Repair
MeSH Terms: conditions — Prostatic Neoplasms | interventions — talazoparib; enzalutamide

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Talazoparib plus enzalutamide
  Interventions: Drug: talazoparib plus enzalutamide
- Arm 2 (Active Comparator): Placebo plus enzalutamide
  Interventions: Drug: Placebo plus enzalutamide

INTERVENTIONS:
Drug: talazoparib plus enzalutamide — experimental arm
  Other Names: Combination arm
  Arms: Arm 1
Drug: Placebo plus enzalutamide — Active comparator arm
  Other Names: Monotherapy arm
  Arms: Arm 2

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of talazoparib in combination with enzalutamide compared with placebo in combination with enzalutamide in participants with DDR-deficient mCSPC.

DETAILED DESCRIPTION:
The study will have 5 periods: prescreening, screening, double-blind treatment, safety follow-up, and long-term follow-up.

Approximately 550 men with mCSPC will be randomized. Eligible participants will be randomly assigned to either of 2 treatment groups as follows:

* Talazoparib in combination with enzalutamide.
* Placebo capsules identical in appearance to talazoparib capsules in combination with enzalutamide.

Talazoparib or identical placebo treatment will be blinded. Enzalutamide (160 mg/day) will be open label. The dose of talazoparib/placebo to be given in combination with enzalutamide is 0.5 mg once daily. Participants with moderate renal impairment (eGFR 30-59 mL/min/1.73 m2 by the MDRD equation) at screening may be enrolled and the talazoparib/placebo dose will be 0.35 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants at least 18 years of age at screening (20 years for Japan, 19 years for Republic of Korea).
2. Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, small cell or signet cell features. If the participant does not have a prior histological diagnosis, a baseline de novo biopsy must be used to confirm the diagnosis and may also be used to support biomarker analysis.
3. Confirmation of DDR gene mutation status by prospective or historical analysis (with sponsor pre-approval) of blood (liquid biopsy) and/or de novo or archival tumor tissue using FoundationOne Liquid CDx or FoundationOne CDx.
4. Willing to provide tumor tissue when available (de novo or archived) for retrospective molecular profiling analysis, if not already provided as part of inclusion criterion 3.
5. Unless prohibited by local regulations or ethics committee decision, consent to a saliva sample collection for retrospective sequencing of the same DDR genes tested on tumor tissue and blood (liquid biopsy), or a subset thereof, and to serve as a germline control in identifying tumor mutations.
6. Ongoing ADT with a GnRH agonist or antagonist for participants who have not undergone bilateral orchiectomy must be initiated before randomization and must continue throughout the study.
7. Metastatic prostate cancer documented by positive bone scan (for bone disease) or metastatic lesions on CT or MRI scan (for soft tissue). Participants whose disease spread is limited to regional pelvic lymph nodes are not eligible. Note: a finding of superscan at baseline is exclusionary.
8. Prior treatment of mCSPC with docetaxel is not permitted.
9. Treatment with estrogens, cyproterone acetate, or first-generation anti-androgens is allowed until randomization.
10. Other prior therapy allowed for mCSPC; ≤3 months of ADT (chemical or surgical) with or without approved NHT in mCSPC (ie, abiraterone + prednisone, apalutamide, or enzalutamide), if required prior to randomization, with no radiographic evidence of disease progression or rising PSA levels prior to Day 1.
11. Participant may have received palliative radiation or surgery for symptomatic control secondary to prostate cancer, which should have been completed at least 2 weeks prior to randomization. NOTE: Radical prostatectomy or definitive radiotherapy to the primary tumor for metastatic castration-sensitive prostate cancer with curative intent is not permitted.
12. ECOG performance status 0 or 1.
13. Adequate organ function within 28 days before the first study treatment on Day 1, defined by the following:

    * ANC ≥1500/µL, platelets ≥100,000/µL, or hemoglobin ≥9 g/dL (may not have received growth factors or blood transfusions within 14 days before obtaining the hematology laboratory tests at screening).
    * Total serum bilirubin <1.5 × ULN (<3 × ULN for participants with documented Gilbert syndrome or for whom indirect bilirubin concentrations suggest an extrahepatic source of elevation).
    * AST or ALT <2.5 × ULN (<5 × ULN if liver function abnormalities are due to hepatic metastasis).
    * Albumin >2.8 g/dL.
    * eGFR ≥30 mL/min/1.73 m2 by the MDRD equation.
14. Sexually active participants that in the opinion of the investigator are capable of ejaculating, must agree to use a condom when having sex with a partner (female or male) from the time of the first dose of study treatment through 4 months after last dose of study treatment (or, if talazoparib/placebo has been stopped more than a month earlier than enzalutamide, through 3 months after last dose of enzalutamide). Must also agree for female partner of childbearing potential to use an additional highly effective form of contraception from the time of the first dose of study treatment through 4 months after last dose of study treatment (or, if talazoparib / placebo has been stopped more than a month earlier than enzalutamide, through 3 months after last dose of enzalutamide) when having sex.
15. Must agree not to donate sperm from the first dose of study treatment to 4 months after the last dose of study treatment (or, if talazoparib/placebo has been stopped more than a month earlier than enzalutamide, through 3 months after last dose of enzalutamide).
16. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures, including being able to manage electronic diaries. The PRO assessments are not required to be completed if a patient does not understand the language(s) available for a specific questionnaire and/or cannot complete the specific questionnaire independently.
17. Capable of giving signed informed consent.
18. For France only: Participants affiliated with the social security system or beneficiaries of an equivalent system.

Exclusion Criteria:

1. Other acute or chronic medical (concurrent disease, infection, including chronic stable HIV, HBV, or HCV infection, or co-morbidity) or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that interferes with a participant's ability to participate in the study, may increase the risk of associated with study participation or study treatment administration, or may interfere with the interpretation of study results, and, in the investigator's judgment, make the participant inappropriate for entry into the study. HIV/HBV/HCV testing is not required unless mandated by local health authority.
2. History of seizure or any condition (as assessed by investigator) that may predispose to seizure (eg, prior cortical stroke, significant brain trauma), including any history of loss of consciousness or transient ischemic attack within 12 months of randomization.
3. Major surgery (as defined by the investigator) within 4 weeks before randomization.
4. Known or suspected brain metastasis or active leptomeningeal disease.
5. Symptomatic or impending spinal cord compression or cauda equina syndrome.
6. Any history of MDS, AML, or prior malignancy except for the following:

   * Carcinoma in situ or non-melanoma skin cancer.
   * A cancer diagnosed and treated ≥3 years before randomization with no subsequent evidence of recurrence.
   * American Joint Committee on Cancer Stage 0 or Stage 1 cancer <3 years before randomization that has a remote probability of recurrence in the opinion of the investigator and the sponsor.
7. In the opinion of the investigator, any clinically significant gastrointestinal disorder affecting absorption.
8. Clinically significant cardiovascular disease, including any of the following:

   * Myocardial infarction or symptomatic cardiac ischemia within 6 months before randomization.
   * Congestive heart failure New York Heart Association class III or IV.
   * History of clinically significant ventricular arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsade de pointes) within 1 year before screening.
   * History of Mobitz II second degree or third-degree heart block unless a permanent pacemaker is in place.
   * Hypotension as indicated by systolic blood pressure <86 mm Hg at screening.
   * Bradycardia as indicated by a heart rate of <45 beats per minute on the screening electrocardiogram.
   * Uncontrolled hypertension as indicated by systolic blood pressure >170 mm Hg or diastolic blood pressure >105 mm Hg at screening. However, participants can be rescreened after adequate control of blood pressure is achieved.
9. Active COVID-19 infection detected by viral test or based on clinical diagnosis (as assessed by investigator). Asymptomatic participants with no active COVID-19 infection detected but positive antibody tests, indicating past infection are allowed.
10. Prior ADT in the adjuvant/neoadjuvant setting, where the completion of ADT was less than 12 months prior to randomization and the total duration of ADT exceeded 36 months.
11. Participant received treatment with systemic glucocorticoids greater than the equivalent of 10 mg per day of prednisone within 4 weeks prior to randomization, intended for the treatment of prostate cancer.
12. Any previous treatment with DNA-damaging cytotoxic chemotherapy (ie, platinum based therapy) within 5 years prior to randomization, except for indications other than prostate cancer.
13. Prior treatment with a PARPi, or known or possible hypersensitivity to enzalutamide, any of enzalutamide capsule excipients or to any talazoparib/placebo capsule excipients.
14. Prior treatment in any setting with NHT, except as described in Inclusion Criterion #10.
15. Current use of potent P-gp inhibitors within 7 days prior to randomization.
16. Treatment with any investigational study intervention within 4 weeks before randomization. Exception: COVID-19 vaccines authorized under an emergency use authorization (or equivalent) can be administered without a washout period.
17. Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF interval >470 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >470 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTc exceeds 470 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
18. Investigator site staff or Sponsor employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
19. For France only: Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric care, as well as adults subject to a legal protection measure (guardianship, curatorship, and safeguard of justice) covered by Articles 1121-6 to 1121-8 of the Public Health Code.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 599 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
radiological Progression-Free Survival | randomization up to 3 years
  time from the date of randomization to first objective evidence of radiographic progression or death, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival | randomization up to 4 years
  time from randomization to death from any cause
Objective response in measurable soft tissue disease | randomization up to 3 years
  proportion of patients with measurable soft tissue disease at baseline with objective response per RECIST 1.1
Duration of response in measurable soft tissue disease | randomization up to 3 years
  duration of responses in patients with measurable soft tissue disease at baseline per RECIST 1.1
Prostate Specific Antigen (PSA) response | randomization up to 3 years
  proportion of patients with PSA response grater than or equal to 50%
Time to PSA progression | randomization up to 3 years
  time from baseline to PSA progression
Time to initiation of antineoplastic therapy | randomization up to 3 years
  Time from randomization to initiation of antineoplastic therapy
Time to first symptomatic skeletal event | randomization up to 3 years
  time from randomization to first symptomatic skeletal event (symptomatic fractures, spinal cord compression, surgery or radiation to the bone whichever is first)
Opiate use for prostate cancer pain | randomization up to 3 years
  time from randomization to opiate use for prostate cancer pain
Incidence of adverse events | randomization up to 3 years
  AEs and SAEs incidence by type and severity (graded by NCI CTCAE version 4.03)
Pharmacokinetic assessment of talazoparib | Weeks 5, 9, 13, and 17
  plasma concentrations of talazoparib
Pharmacokinetic assessment of enzalutamide and its metabolite | Weeks 5, 9, 13, and 17
  plasma concentrations of enzalutamide and its metabolite
Relationship between ctDNA burden and outcome | randomization up to 3 years
  ctDNA burden at baseline and on study
Patient-reported outcomes in pain symptoms - change from baseline | randomization up to 3 years
  change from baseline in patient-reported pain symptoms per Brief Pain Inventory Short Form (BPI-SF)
Patient-reported outcomes in pain symptoms - time to deterioration | randomization up to 3 years
  time to deterioration in patient-reported pain symptoms per Brief Pain Inventory Short Form (BPI-SF)
Patient-reported outcomes in cancer specific general health status - change from baseline | randomization up to 3 years
  change from baseline in participant-reported general health status per EQ-5D-5L
Patient-reported outcomes in cancer specific global health status/QoL - change from baseline | randomization up to 3 years
  change from baseline in patient-reported Global health status/QoL per EORTC QLQ-C30
Patient-reported outcomes in cancer specific global health status/QoL - time to definitive deterioration | randomization up to 3 years
  time to definitive deterioration in patient-reported global health status/QoL per EORTC QLQ-C30
Patient-reported outcomes in cancer specific symptoms - time to definitive deterioration | randomization up to 3 years
  time to definitive deterioration in disease specific urinary symptoms per EORTC QLQ-PR25
Patient-reported outcome: cancer specific functioning, and symptoms - change from baseline | randomization up to 3 years
  change from baseline in PGI-S

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (306):
- United States (43):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Institute of Urology, PLLC, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Adventist Health Glendale, Glendale, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth, Orlando, Florida
  - AdventHealth Medical Group Hematology and Oncology, Orlando, Florida
  - Investigational Drug Services, Advent Health Orlando, Orlando, Florida
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Austell, Georgia
  - Wellstar Cobb Hospital, Austell, Georgia
  - Northwest Georgia Oncology Centers, a Service of Tanner Medical Center Villa Rica, Carrollton, Georgia
  - West Georgia Infusion Center, a Service of Tanner Medical Center Villa Rica, Carrollton, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Cartersville, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Douglasville, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - Comprehensive Urologic Care, SC, Lake Barrington, Illinois
  - Mid-Illinois Hematology & Oncology Associates, Ltd, Normal, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Revive Research Institute, Inc., Farmington Hills, Michigan
  - David C. Pratt Cancer Center, St Louis, Missouri
  - New Jersey Cancer Care, P.A., Belleville, New Jersey
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Indian Path Community Hospital, Kingsport, Tennessee
  - Kelsey Research Foundation, Houston, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - oncology Consultants, P.A., Houston, Texas
  - Houston Metro Urology, Houston, Texas
  - Oncology Consultants P.A., Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Texas Oncology-Deke Slayton Cancer Center, Webster, Texas
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah
- Argentina (7):
  - COIBA, Berazategui, Buenos Aires
  - Centro de Investigacion Pergamino SA - Clinica Pergamino SA, Pergamino, Buenos Aires
  - Centro de Investigaciones Clínicas - Clínica Viedma, Viedma, Río Negro Province
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Centro Oncologico Korben, Caba
  - Instituto Médico Especializado Alexander Fleming, CABA
  - Centro Medico Privado CEMAIC, Córdoba
- Australia (9):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Cancer Care Wollongong Pty Limited, Wollongong, New South Wales
  - Gallipoli Medical Research Foundation, Greenslopes Private Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Epworth Freemasons-Epworth HealthCare, East Melbourne, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Epworth Foundation Trading as Epworth HealthCare, Richmond, Victoria
  - Western Health, Sunshine Hospital, St Albans, Victoria
- Belgium (9):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Anderlecht
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - AZ (Algemeen Ziekenhuis) Maria Middelares, Ghent
  - AZ (Algemeen Ziekenhuis) Sint-Lucas, Ghent
  - AZ (Algemeen Ziekenhuis) Groeninge, Kortrijk
  - CHU de Liege, Liège
  - ZNA Jan Palfijn, Merksem
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagyurishte
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Independent medical-diagnostic laboratory "Medisken" EOOD, Plovdiv
  - Complex Oncology Center - Shumen EOOD, Shumen
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
  - Complex Oncology Center - Stara Zagora Ltd., Stara Zagora
  - MRI SMDLOD "Mediscan" Ltd, Stara Zagora
  - UMHAT "Prof. Dr. Stoyan Kirkovich", Stara Zagora
- Canada (13):
  - Prostate Cancer Centre, Calgary, Alberta
  - Centre of Applied Urology Research, Nova Scotia Health Authority, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Organisation Lawson Health Research Institute, London, Ontario
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - University Health Network-Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre integre universitaire de sante et de services sociaux Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Urology South Shore Research, Greenfield Park, Quebec
  - Centre Hospitalier de I'Universite de Montreal (CHUM), Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- China (25):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Lanzhou university second hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - The First hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The first affiliated hospital of Ningbo university, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The First Affiliated Hospital Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
- Czechia (5):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
  - Fakultni nemocnice Bulovka, Praha 8- Liben
- Finland (6):
  - Helsinki University Hospital, Helsinki
  - Docrates Cancer Center, Helsinki
  - Clinical Research Institute Helsinki University Central Hospital Ltd, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (15):
  - CHU Morvan de Brest, Brest, Brittany Region
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Clinique Belharra, Bayonne
  - Hopital Prive le Bois, Lille
  - Centre Leon Berard, Lyon
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - Clinique La Croix du Sud - Ramsay Sante, Quint-Fonsegrives
  - Institut Jean Godinot, Reims
  - CHP Saint-Grégoire, Saint-Grégoire
  - Hopitaux Universitaires de Strasbourg - ICANS (Institut de Cancerologie Strasbourg Europe), Strasbourg
  - Institut de cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
  - Hopital Henri Mondor, Créteil, Île-de-France Region
- Germany (11):
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Urologische Gemeinschaftspraxis Wesel, Wesel, North Rhine-Westphalia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charite Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Urologicum Duisburg, Duisburg
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Institut fuer Diagnostische und Interventionelle Radiologie, Göttingen
  - Universitaetsklinik Heidelberg, Heidelberg
  - Uro-/Onkologisches Zentrum, Leipzig
  - Studienpraxis Urologie, Nürtingen
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (4):
  - Péterfy Kórház-Rendelőintézet és Manninger Jenő Országos Traumatológiai Intézet, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
- India (12):
  - Gujarat Hospital - Gastro and Vascular Centre, Surat, Gujarat
  - Artemis hospital, Gurugram, Haryana
  - Medanta- The Medicity hospital, Gurugram, Haryana
  - Bhaktivedanta Hospital and Research Institute, Mumbai, Maharashtra
  - Sahyadri Clinical Research & Development Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Sahyadri Hospitals Private Limited, Pune, Maharashtra
  - Indraprastha Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute and Research Centre, New Delhi, National Capital Territory of Delhi
  - Valentis Cancer Hospital, Meerut, Uttar Pradesh
  - Netaji Subhas Chandra Bose Cancer Hospital, Kolkata, West Bengal
  - Indraprastha Apollo Hospitals, New Delhi
- Italy (15):
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola Malpighi, Bologna, BO
  - ASST Cremona, Cremona, CR
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" (IRST), Meldola, FC
  - Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale - Napoli, Napoli, Naples
  - Centro di Riferimento Oncologico di Aviano (CRO) IRCCS, Aviano, PN
  - Ospedale Santa Chiara, Trento, TN
  - AOU San Luigi Gonzaga, Orbassano, TO
  - Azienda Provinciale per i Servizi Sanitari, della Provincia Autonoma di Trento, Trento, Trentino-Alto Adige
  - Azienda Unita Sanitaria Locale Toscana Sud-Est, Arezzo
  - Ospedale San Donato, Arezzo
  - IRCCS Istituto Tumori "Giovanni Paolo II" di Bari, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - ASST degli Spedali Civili de Brescia, Brescia
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (22):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University School of Medicine & Hospital, Hirosaki, Aomori
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokosukakyosai, Yokosuka, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku, Tokyo
  - Keio university hospital, Shinjuku-ku, Tokyo
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Tokushima University Hospital, Tokushima
  - Yamagata University Hospital, Yamagata
- Mexico (7):
  - Preparaciones Oncológicas S.C., León, Guanajuato
  - Axis Heilsa S. de R.L. de C.V., Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - Oncologia Integral Satelite SA de CV, Naucalpan, State of Mexico
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
- Netherlands (2):
  - Meander Medisch Centrum, Amersfoort, Utrecht
  - Stichting HagaZiekenhuis, The Hague
- Sykehuset Innlandet Gjoevik, Gjøvik, Norway
- Russia (16):
  - MRRC n.a. A.F. Tsyb - branch of FSBI "NMRC of Radiology" Minzdrav Russia, Obninsk, Kaluga Oblast
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - Limited Liability Company "4D Ultrasound Clinic" (LLC "4D Ultrasound Clinic"), Pyatigorsk, Stavropol Kray
  - Evimed Llc, Chelyabinsk
  - SBIH "Chelyabinsk Regional Clinical Centre of Oncology and Nuclear Medicine", Chelyabinsk
  - Regional Budgetary Healthcare Institution "Ivanovskiy Regional Oncology Dispensary" (RBHI "IvROD"), Ivanovo
  - Federal State Budgetary Institution "Russian Research Center of Roentgenology and Radiology" of the, Moscow
  - Branch of the Limited Liability Company "Hadassah Medical Ltd.", Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with ambulance", Moscow
  - BHI of Omsk region "Clinical Oncological Dispensary", Omsk
  - LLC "Medicina Severnoy Stolitsy", Saint Petersburg
  - LLC "Severo-Zapadny Medical Center", Saint Petersburg
  - Private Institution Educational Organization of Higher Education "Medical University "REAVIZ", Samara
  - SAHI Republican Clinical Oncology Dispensary under the Ministry of Health, Republic of Bashkortostan, Ufa
  - Budgetary Healthcare Institution of Vologda region "Vologda Regional Clinical Hospital", Vologda
  - State Budgetary Institution of Healthcare of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl
- Slovakia (7):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - Narodny onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - UROEXAM, spol. s r.o., Nitra
  - POKO Poprad s.r.o., Poprad
  - MILAB s.r.o., Prešov
  - Privatna urologicka ambulancia, s.r.o., Trenčín
- South Africa (6):
  - 15 Eton Road, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - WCR Office, Johannesburg, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd, Johannesburg, Gauteng
  - Wits Clinical Research, Parktown, Gauteng
  - Clinical Research Unit, University of Pretoria, Pretoria, Gauteng
- South Korea (11):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (18):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Institut Català d'Oncologia de l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Comunidad de
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Fundación Instituto Valenciano de Oncología, Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Politecnic Universitari La Fe, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Turkey (Türkiye) (7):
  - Adana City Training and Research Hospital, Adana
  - Ankara University Faculty of Medicine, Ankara
  - Ankara City Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul University, Cerrahpasa Faculty of Medicine, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Inonu University, Faculty of Medicine, Malatya
- Ukraine (9):
  - MI Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council; Chemotherapy Department, Kryviy Rih, Dnipropetrovsk Oblast
  - Medical & diagnostic center of LISOD-Israeli Oncological Hosp "MedX-ray International Group", Pliuty Village, Kyiv Oblast
  - Asklepion Medical Center, Khodosovka, Kyivska Oblast
  - National Cancer Institute, Kyiv, Kyivska Oblast
  - Municipal Ent "Dnipropetrovsk Regional Clinical Hosp (I.I.Mechnikov Dnipropetrovsk Regional council), Dnipro
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, Dnipro
  - Municipal Non-Commercial Enterprise of Kharkiv Regional Council Regional Medical Clinical Center of, Kharkiv
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Kharkiv
  - Comm Noncommerc Entp Lviv Reg Council "Lviv Oncological Regional Therapeutical and Diagnostic Cntre, Lviv
- United Kingdom (11):
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone, KENT
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire
  - NHS Lothian, Edinburgh, Midlothian
  - Greater Glasgow Health Board J B Russell House, Gartnavel Royal Hospital, Glasgow, Scotland
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Agarwal N, Saad F, Azad AA, Mateo J, Matsubara N, Shore ND, Chakrabarti J, Chen HC, Lanzalone S, Niyazov A, Fizazi K. TALAPRO-3 clinical trial protocol: phase III study of talazoparib plus enzalutamide in metastatic castration-sensitive prostate cancer. Future Oncol. 2024 Mar;20(9):493-505. doi: 10.2217/fon-2023-0526. Epub 2023 Oct 26. PMID 37882449
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441052